CLINICAL TRIAL: NCT02542254
Title: A Phase II, Randomised, Double Blind, Placebo Controlled, Six Way Crossover Study to Assess the Bronchodilator Effect of RPL554 Administered on Top of Salbutamol and Ipratropium in Patients With COPD.
Brief Title: The Effects of RPL554 on Top of Standard COPD Reliever Medications
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Verona Pharma plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RPL554-009-2015; 2015-002536-41 (EudraCT Number)
Record Dates: First submitted 2015-08-30; First posted 2015-09-04 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol; Ipratropium; ensifentrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Salbutamol alone (Active Comparator): 200 micrograms salbutamol, ipratropium matched placebo and RPL554 matched placebo
  Interventions: Drug: Salbutamol; Drug: Ipratropium matched placebo; Drug: RPL554 matched placebo
- Salbutamol and RPL554 (Experimental): 200 micrograms salbutamol, ipratropium matched placebo and 6 mg RPL554
  Interventions: Drug: Salbutamol; Drug: RPL554; Drug: Ipratropium matched placebo
- Ipratropium (Active Comparator): Salbutamol matched placebo, 40 micrograms ipratropium and RPL554 matched placebo
  Interventions: Drug: Ipratropium; Drug: Salbutamol matched placebo; Drug: RPL554 matched placebo
- Ipratropium and RPL554 (Experimental): Salbutamol matched placebo, 40 micrograms ipratropium and 6 mg RPL554
  Interventions: Drug: Ipratropium; Drug: RPL554; Drug: Salbutamol matched placebo
- RPL554 (Experimental): Salbutamol matched placebo, ipratropium matched placebo and 6 mg RPL554
  Interventions: Drug: RPL554; Drug: Salbutamol matched placebo; Drug: Ipratropium matched placebo
- Placebo (Placebo Comparator): Salbutamol matched placebo, ipratropium matched placebo and RPL554 matched placebo
  Interventions: Drug: Salbutamol matched placebo; Drug: Ipratropium matched placebo; Drug: RPL554 matched placebo

INTERVENTIONS:
Drug: Salbutamol — 200 micrograms salbutamol administered using a pressurised metered dose inhaler (pMDI)
  Arms: Salbutamol alone; Salbutamol and RPL554
Drug: Ipratropium — 40 micrograms ipratropium administered using a pMDI
  Arms: Ipratropium; Ipratropium and RPL554
Drug: RPL554 — 6 mg RPL554 administered using a nebuliser
  Arms: Ipratropium and RPL554; RPL554; Salbutamol and RPL554
Drug: Salbutamol matched placebo — Placebo pMDI
  Arms: Ipratropium; Ipratropium and RPL554; Placebo; RPL554
Drug: Ipratropium matched placebo — Placebo pMDI
  Arms: Placebo; RPL554; Salbutamol alone; Salbutamol and RPL554
Drug: RPL554 matched placebo — Nebulised placebo
  Arms: Ipratropium; Placebo; Salbutamol alone

SUMMARY:
This study evaluates the addition of RPL554 to standard reliever medications for chronic obstructive pulmonary disorder (COPD). All patients will receive the same six treatments in a randomised sequence:

1. salbutamol,
2. ipratropium,
3. salbutamol + RPL554,
4. ipratropium + RPL554,
5. RPL554
6. Placebo

DETAILED DESCRIPTION:
The purpose of this study is to investigate if RPL554 has an additive bronchodilator effect when administered in combination with standard of care bronchodilators in patients with COPD.This study investigates the pharmacodynamic effect of RPL554 using spirometry and whole body plethysmography compared to placebo, when administered in addition to a beta2 agonist (salbutamol), a muscarinic antagonist (ipratropium) or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* Males not donating sperm and using adequate contraception or females who are surgically sterile or postmenopausal
* 12-lead ECG showing:Heart rate 45 to 90 bpm, QTcF≤450 msec, QRS ≤120 msec, PR interval ≤220 msec, no clinically significant abnormality
* Capable of complying with all study restrictions and procedures including ability to use the study nebuliser correctly.
* BMI 18 to 33 kg/m2 with a minimum weight of 45 kg.
* COPD diagnosis for at least 1 year and clinically stable COPD in previous 4 weeks
* Demonstrates reversibility to bronchodilator (two puffs of salbutamol followed by two puffs of ipratropium) via spirometry:

  * Post-bronchodilator FEV1/forced vital capacity (FVC) ratio of ≤0.70
  * Post-bronchodilator FEV1 ≥40 % and ≤80% of predicted normal
  * ≥150 mL increase from pre-bronchodilator FEV1
* Chest X-ray showing no abnormalities
* Meet the concomitant medication restrictions and be expected to do so for the rest of the study.
* Smoking history of ≥10 pack years.
* Capable of withdrawing from long acting bronchodilators throughout the study and short acting bronchodilators for 8 hours prior to study treatment.

Exclusion Criteria:

* History of life-threatening COPD including Intensive Care Unit admission and/or requiring intubation.
* COPD exacerbation requiring oral steroids in the previous 3 months
* History of one or more hospitalisations for COPD in the previous 12 months
* Respiratory tract infection (both upper and lower) treated with antibiotics in previous 12 weeks
* Evidence of cor pulmonale or clinically significant pulmonary hypertension.
* Other respiratory disorders
* Previous lung resection or lung reduction surgery.
* Oral therapies for COPD in the previous 3 months and throughout the study.
* Drug or alcohol abuse in the past 3 years
* Received an experimental drug within 3 months or five half lives, whichever is longer.
* Prior exposure to RPL554
* Patients with a history of chronic uncontrolled disease that the Investigator believes are clinically significant.
* Documented cardiovascular disease in last 3 months
* Major surgery, (requiring general anaesthesia) in the previous 6 weeks, or will not have fully recovered from surgery, or planned surgery through the end of the study.
* History of malignancy of any organ system within 5 years with the exception of localised skin cancers (basal or squamous cell)
* Clinically significant abnormal values for safety laboratory tests
* A disclosed history, or one known to the Investigator, of significant non compliance in previous investigational studies or with prescribed medications.
* Requires oxygen therapy, even on an occasional basis.
* Inability to adequately perform whole body plethysmography.
* Any other reason that the Investigator considers makes the subject unsuitable to participate.
* Patients with known hypersensitivity to atropine or its derivatives, or to ipratropium bromide, salbutamol or RPL554 or their excipients/components.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
8 hour spirometry | 8 hours
  Forced expired volume in one second (FEV1) over 8 hours post-dose

SECONDARY OUTCOMES:
12 hour spirometry | 12 hours
  FEV1 over 4, 6 and 12 hours post-dose
Whole body plethysmography | 4 hours
  Functional residual capacity, residual volume, total lung capacity, specific airway conductance, specific airway resistance at 1 and 4 hours post-dose
Area under the curve (AUC) | 12 hours
  AUC for RPL554 plasma concentration
Maximum plasma concentration (Cmax) | 12 hours
  Cmax for RPL554 plasma concentration
Time to maximum plasma concentration (Tmax) | 12 hours
  Tmax for RPL554 plasma concentration
Adverse events | Up to 94 days
  Continuous measurement of adverse events throughout the study
Safety laboratory tests | Up to 94 days
  Laboratory safety tests at screening, before each treatment and end of study
ECG | Up to 94 days
  12 lead ECG at screening, before and up to 12 hours after each treatment and end of study
Vital signs | Up to 94 days
  Blood pressure and pulse rate at screening, before and up to 12 hours after each treatment and end of study

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, Principal Investigator — Medicines Evaluation Unit
Locations (1):
- Medicines Evaluation Unit, Manchester, United Kingdom

REFERENCES:
- [Derived] Singh D, Abbott-Banner K, Bengtsson T, Newman K. The short-term bronchodilator effects of the dual phosphodiesterase 3 and 4 inhibitor RPL554 in COPD. Eur Respir J. 2018 Nov 1;52(5):1801074. doi: 10.1183/13993003.01074-2018. Print 2018 Nov. PMID 30166326